CLINICAL TRIAL: NCT00615706
Title: Study to Evaluate the Impact of Obesity on Airway Inflammation and Mechanics in Asthmatics
Acronym: ABI/BALA
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Critical Therapeutics (Industry)
Responsible Party: Fernando Holguin, MD, MPH, Emory University
Other Study IDs: 345-2004; Emory IRB ID 345-2004
Record Dates: First submitted 2008-02-04; First posted 2008-02-14 (Estimated); Last update posted 2008-09-23 (Estimated); Status verified 2008-09

CONDITIONS: Asthma
Keywords: asthma, inhaled corticosteroids
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, urine, DNA, exhaled breath condensate. For substudy participants, bronchoalveolar lavage samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Asthmatics
  Interventions: Other: No intervention
- 2: Healthy volunteers (without asthma)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — no intervention

SUMMARY:
In the United States there has been a dramatic increase in the number of people who are obese and in the number of people who have asthma. Both are considered serious public health concerns. Several studies have shown that becoming obese or overweight can increase the risk of developing asthma or can make asthma symptoms more severe and difficult to control. How obesity affects asthma is not fully understood. This research study will examine whether obesity affects the amount of inflammation that is present in the lungs of people with asthma, and will also examine whether obesity leads to narrow and stiff airways.

Participation in this study involves 2 visits in order to complete questionnaires, various pulmonary function tests, as well as the collection of blood, urine, and exhaled breath condensate specimens.

This research study includes optional genetic and bronchoscopy substudies.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 70 years of age
* If asthmatic, currently taking a short acting beta agonist and an inhaled corticosteroid
* Never smoked or limited smoking history

Exclusion Criteria:

* Current upper respiratory illness (other than asthma)
* Illegal drug use within past month
* Consumption of more than 6 alcoholic drinks per week
* Active, pronounced rhinitis or sinusitis
* Pregnancy
* Currently taking oral steroids or steroid injection over the past month
* Asthma exacerbation over the past month
* Certain medical illnesses

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asthmatics and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2005-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Emory Crawford Long Hospital, Clinical Research Center, Atlanta, Georgia, United States